CLINICAL TRIAL: NCT00003622
Title: Phase II Study of Vinorelbine With Paclitaxel in the Treatment of Hormone-Refractory Prostate Cancer
Brief Title: Vinorelbine Plus Paclitaxel in Treating Patients With Metastatic Prostate Cancer That Is Refractory to Hormone Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: James Ahlgren (Other)
Responsible Party: Sponsor-Investigator, James Ahlgren, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCC-4097; CDR0000066701 (Registry Identifier: PDQ (Physician Data Query)); GW-GWCC-4097; NCI-V98-1486
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Paclitaxel; Vinorelbine

ARMS (1):
- paclitaxel + vinorelbine (Experimental)
  Interventions: Drug: paclitaxel; Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: paclitaxel
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine plus paclitaxel in treating patients with metastatic prostate cancer that is refractory to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical benefit response (including improvement in quality of life) of vinorelbine and paclitaxel in patients with metastatic hormone-refractory prostate cancer. II. Correlate PSA response with clinical benefit response in these patients. III. Determine the objective response rate and duration of remission in patients with measurable disease treated with this regimen. IV. Further assess the toxicity of this combination in a cohort of prostate cancer patients. V. Examine the survival characteristics of these patients undergoing this regimen.

OUTLINE: This an open label study. Patients receive vinorelbine IV over 6-10 minutes on days 1, 2, and 3 and paclitaxel IV over 3 hours on day 3 following vinorelbine. Course repeats every 28 days in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before each treatment course. Patients are followed until death.

PROJECTED ACCRUAL: A total of 30 patients will be accrued into this study over 15-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the prostate that is hormone refractory Hormone-refractory defined as at least 50% increase in PSA while continuing hormonal therapy Must have received prior hormonal manipulation including either orchiectomy or LHRH agonist Must be symptomatic and on a stable dose of pain medication No documented CNS involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 1-2 Life expectancy: At least 16 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.8 mg/dL Renal: Creatinine no greater than 1.8 mg/dL Other: Not HIV positive No concurrent infection No concurrent medical or psychiatric illness that precludes study compliance No prior or concurrent second malignancy in the past 5 years except basal or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 4 weeks since prior antiandrogens If patients have received prior antiandrogens, PSA levels are reassessed at 4 week intervals until there is no decrease in PSA levels before registration into this study Radiotherapy: Prior radiotherapy allowed Must have recovered from prior radiotherapy Concurrent radiotherapy for symptomatic bone lesion allowed Surgery: Not specified Other: No other concurrent therapeutic study

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-01; Primary Completion 2008-05 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Ahlgren, MD, Study Chair — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States